CLINICAL TRIAL: NCT03409614
Title: A Two-Part Randomized, Phase 3 Study of Combinations of Cemiplimab (Anti-PD-1 Antibody) and Platinum-based Doublet Chemotherapy in First-line Treatment of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Combinations of Cemiplimab (Anti-PD-1 Antibody) and Platinum-based Doublet Chemotherapy in Patients With Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2810-ONC-16113; 2017-001311-36 (EudraCT Number)
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage IIIB; Stage IIIC; Stage IV; Non-squamous NSCLC; Squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: Open label Part 2: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Chemo (Other): Part 1: Chemotherapy
  Interventions: Other: Chemotherapy; Drug: Placebo
- REGN2810+Chemo Part 1 (Experimental): Part 1: REGN2810+chemo
  Interventions: Drug: REGN2810
- REGN2810+AbbrevChemo+ipi (Experimental): Part 1: REGN2810+abbrev chemo+ipi
  Interventions: Drug: REGN2810/chemo/ipi
- Placebo+Chemo (Experimental): Part 2: Placebo plus chemo
  Interventions: Drug: Placebo
- REGN2810+Chemo Part 2 (Experimental): Part 2: REGN2810+chemo
  Interventions: Drug: REGN2810

INTERVENTIONS:
Drug: REGN2810 — REGN2810 plus Platinum-based doublet chemotherapy Part 1 and Part 2
  Other Names: cemiplimab
  Arms: REGN2810+Chemo Part 1; REGN2810+Chemo Part 2
Drug: REGN2810/chemo/ipi — REGN2810 plus abbreviated chemotherapy plus Ipilimumab Part 1
  Other Names: cemiplimab
  Arms: REGN2810+AbbrevChemo+ipi
Other: Chemotherapy — Platinum-based doublet chemotherapy Part 1
  Arms: Chemo
Drug: Placebo — Matching placebo Part 2
  Arms: Chemo; Placebo+Chemo

SUMMARY:
The primary objectives of this study are:

Part 1: To compare the overall survival (OS) of cemiplimab/chemo-f and cemiplimab/chemo-l/ipi versus platinum-based doublet chemotherapy in the first-line treatment of patients with advanced squamous or nonsquamous non-small cell lung cancer (NSCLC) with tumors expressing PD-L1 in <50% of tumor cells.

Part 2: To compare the OS of cemiplimab/chemo-f with placebo/chemo-f in the first-line treatment of patients with advanced squamous or non-squamous NSCLC irrespective of PD-L1 expression.

The key secondary objectives are:

Part 1: To compare the progression-free survival (PFS) and objective response rate (ORR) of cemiplimab/chemo-f and cemiplimab/chemo-l/ipi versus chemo-f in the first-line treatment of patients with advanced squamous or non-squamous NSCLC and tumors expressing PD-L1 in <50% of tumor cells.

Part 2: To compare the PFS and ORR of cemiplimab/chemo-f versus placebo/chemo-f in the first-line treatment of patients with advanced squamous or non-squamous NSCLC irrespective of PD-L1 expression.

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women ≥20 years of age for Japanese patients
2. Patients with histologically or cytologically documented squamous or non-squamous NSCLC with stage IIIB or IIIC disease who are not candidates for treatment with definitive concurrent chemoradiation or patients with stage IV disease if they have not received prior systemic treatment for recurrent or metastatic NSCLC
3. Availability of an archival (≤5 months) or on-study obtained formalin-fixed, paraffin-embedded tumor tissue sample from a metastatic or recurrent site, which has not previously been irradiated
4. Part 1 only: Expression of PD-L1 in <50% of tumor cells determined by a commercially available assay performed by the central laboratory
5. At least 1 radiographically measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
7. Anticipated life expectancy of at least 3 months

Key Exclusion Criteria:

1. Part 1 only: Patients who have never smoked, defined as smoking ≤100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression
3. Patients with tumors tested positive for Epidermal growth factor receptor (EGFR) gene mutations, Anaplastic lymphoma kinase (ALK) gene translocations, or C-ros oncogene receptor tyrosine kinase(ROS1) fusions
4. Encephalitis, meningitis, or uncontrolled seizures in the year prior to enrollment
5. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years
6. Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk of immune-related treatment-emergent adverse events (irTEAEs)
7. Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 32 months

SECONDARY OUTCOMES:
Progression-free survival | Up to 32 months
Objective response rate | Up to 32 months
Duration of Response (DOR) | Up to 32 months
Best overall response (BOR) | Up to 32 months
Incidence of Treatment-emergent adverse events (TEAEs) | Up to 32 months
Incidence of Dose-limiting toxicities (DLTs) | Up to 32 months
  Part 1 only
Incidence of serious adverse events (SAEs) | Up to 32 months
Incidence of deaths | Up to 32 months
Incidence of laboratory abnormalities | Up to 32 months
Overall survival rate | 12 months
Overall survival rate | 18 months
Overall survival rate | 24 months
Quality of life as measured by EORTC QLQ-C30 | Up to 32 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Quality of life as measured by EORTC QLQ-LC13 | Up to 32 months
  Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (114):
- United States (9):
  - Regeneron Research Site, Rancho Mirage, California
  - Regeneron Research Site, Riverside, California
  - Regeneron Research Site, Whittier, California
  - Regeneron Research Site, Orange City, Florida
  - Regeneron Research Site, St. Petersburg, Florida
  - Regeneron Research Site, Wichita, Kansas
  - Regeneron Research Site, Bethesda, Maryland
  - Regeneron Research Site, Farmington, New Mexico
  - Regeneron Research Site, Gettysburg, Pennsylvania
- Regeneron Research Site, Vienna, Austria
- China (12):
  - Regeneron Research Site, Baoding
  - Regeneron research Site, Beijing
  - Regeneron Research Site, Changsha
  - Regeneron Research Site, Guangzhou
  - Regeneron Research Site, Hangzhou
  - Regeneron Research Site, Jinan
  - Regeneron Research Site, Linyi
  - Regeneron Research Site, Nanjing
  - Regeneron Research Site, Shanghai
  - Regeneron Research Site, Shenyang
  - Regeneron Research Site, Xiangyang
  - Regeneron Research Site, Zhengzhou
- France (9):
  - Regeneron Research Site, Bayonne
  - Regeneron Research Site, Créteil
  - Regeneron Research Site, Le Mans
  - Regeneron Research Site, Lille
  - Regeneron Research Site, Lyon
  - Regeneron Research Site, Mont-de-Marsan
  - Regeneron Research Site, Saint-Herblain
  - Regeneron Research Site, Saint-Mandé
  - Regeneron Research Site, Strasbourg
- Georgia (4):
  - Regeneron Research Site, Batumi
  - Regeneron Research Site, Tbilisi
  - Regeneron Research Site #1, Tbilisi
  - Regeneron Research Site #2, Tbilisi
- Greece (6):
  - Regeneron Research Site, Thessaloniki, Macedonia
  - Regeneron Research Site, Athens
  - Regeneron Research Site, Kifissia
  - Regeneron Research Site, Larissa
  - Regeneron Research Site, Pylaia
  - Regeneron Research Site, Thessaloniki
- Ireland (2):
  - Regeneron Research Site, Dublin
  - Regeneron Research Site, Limerick
- Italy (8):
  - Regeneron Research Site, Cremona
  - Regeneron Research Site, Meldola
  - Regeneron Research Site, Milan
  - Regeneron Research Site, Monserrato
  - Regeneron Research Site, Piacenza
  - Regeneron Research Site, Saronno
  - Regeneron Research Site, Terni
  - Regeneron Research Site, Treviglio
- Lithuania (2):
  - Regeneron Research Site, Klaipėda
  - Regeneron Research Site, Vilnius
- Malaysia (8):
  - Regeneron Research Site, Kuala Lumpur, Kuala Lumpur
  - Regeneron Research Site, George Town
  - Regeneron Research Site, Johor Bahru
  - Regeneron Research Site, Kota Kinabalu
  - Regeneron Research Site, Kuala Lumpur
  - Regeneron Research Site, Kuantan
  - Regeneron Research Site, Pulau Pinang
  - Regeneron Research Site, Tanjung Bungah
- Poland (9):
  - Regeneron Research Site, Gdynia, Pomeranian Voivodeship
  - Regeneron Research Site, Lodz
  - Regeneron Research Site, Lublin
  - Regeneron Research Site, Olsztyn
  - Regeneron Research Site, Otwock
  - Regeneron Research Site, Poznan
  - Regeneron Research Site, Rzeszów
  - Regeneron Research Site, Torun
  - Regeneron Research Site, Wodzisław Śląski
- Romania (2):
  - Regeneron Research Site, Cluj-Napoca
  - Regeneron Research Site, Craiova
- Russia (18):
  - Regeneron Research Site, Ufa, Republic Bashkortost
  - Regeneron Research Site, Arkhangelsk
  - Regeneron Research Site, Belgorod
  - Regeneron Research Site, Chelyabinsk
  - Regeneron Research Site, Kaluga
  - Regeneron Research Site, Kazan'
  - Regeneron Research Site, Kursk
  - Regeneron Research Site, Moscow
  - Regeneron Research Site, Moscow Region
  - Regeneron Research Site, Omsk
  - Regeneron Research Site, Pushkin
  - Regeneron Research Site, Pyatigorsk
  - Regeneron Research Site, Saint Petersburg
  - Regeneron Research Site, Samara
  - Regeneron Research Site, Saransk
  - Regeneron Research Site, Sochi
  - Regeneron Research Site, Tomsk
  - Regeneron Research Site, Yekaterinburg
- Regeneron Research Site, Banka, Slovakia
- South Korea (6):
  - Regeneron Research Site, Cheongju-si
  - Regeneron Research Site, Incheon
  - Regeneron Research Site, Jeonju
  - Regeneron Research Site, Seongnam-si
  - Regeneron Research Site, Seoul
  - Regeneron Research Site, Suwon
- Thailand (8):
  - Regeneron Research Site #2, Ratchathewi, Bangkok
  - Regeneron Research Site, Muang, Changwat Chiang Rai
  - Regeneron Research Site, A. Mueang, Changwat Lampang
  - Regeneron Research Site, Muang, Changwat Phitsanulok
  - Regeneron Research Site, Hat Yai, Changwat Songkhla
  - Regeneron Research Site, Udon Thani, Udonthani
  - Regeneron Research Site, Muang
  - Regeneron Research Site #1, Ratchathewi
- Turkey (Türkiye) (3):
  - Regeneron Research Site, Adana
  - Regeneron Research Site, Ankara
  - Regeneron Research Site, Istanbul
- Ukraine (6):
  - Regeneron Research Site, Dnipro
  - Regeneron Research Site, Kharkiv
  - Regeneron Research Site, Kiev
  - Regeneron Research Site, Kirovohrad
  - Regeneron Research Site, Uzhhorod
  - Regeneron Research Site, Vinnytsia

REFERENCES:
- [Derived] Zhao B, Qi H, Wu J, Ma W. Cemiplimab Plus Chemotherapy Could Be a First-Line Option for Advanced and Metastatic NSCLC: Results From the Phase 3 EMPOWER-Lung 3 Part 2 Trial. J Thorac Oncol. 2023 Jul;18(7):e72-e73. doi: 10.1016/j.jtho.2023.04.001. No abstract available. PMID 37348996
- [Derived] Makharadze T, Gogishvili M, Melkadze T, Baramidze A, Giorgadze D, Penkov K, Laktionov K, Nemsadze G, Nechaeva M, Rozhkova I, Kalinka E, Li S, Li Y, Kaul M, Quek RGW, Pouliot JF, Seebach F, Lowy I, Gullo G, Rietschel P. Cemiplimab Plus Chemotherapy Versus Chemotherapy Alone in Advanced NSCLC: 2-Year Follow-Up From the Phase 3 EMPOWER-Lung 3 Part 2 Trial. J Thorac Oncol. 2023 Jun;18(6):755-768. doi: 10.1016/j.jtho.2023.03.008. Epub 2023 Mar 29. PMID 37001859
- [Derived] Gogishvili M, Melkadze T, Makharadze T, Giorgadze D, Dvorkin M, Penkov K, Laktionov K, Nemsadze G, Nechaeva M, Rozhkova I, Kalinka E, Gessner C, Moreno-Jaime B, Passalacqua R, Li S, McGuire K, Kaul M, Paccaly A, Quek RGW, Gao B, Seebach F, Weinreich DM, Yancopoulos GD, Lowy I, Gullo G, Rietschel P. Cemiplimab plus chemotherapy versus chemotherapy alone in non-small cell lung cancer: a randomized, controlled, double-blind phase 3 trial. Nat Med. 2022 Nov;28(11):2374-2380. doi: 10.1038/s41591-022-01977-y. Epub 2022 Aug 25. PMID 36008722